CLINICAL TRIAL: NCT06012279
Title: Clinical Outcomes of Dapagliflozin in Acute Heart Failure With Reduced Ejection Fraction, a Randomized Controlled Trial (CODA-HFrEF)
Brief Title: Clinical Outcomes of Dapagliflozin in Acute Heart Failure With Reduced Ejection Fraction (CODA-HFrEF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Aswan Heart Centre (Other)
Responsible Party: Principal Investigator, Hossameldin Elsayed Khalifa Hussein, Assistant Lecturer of Cardiology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-343-2021
Record Dates: First submitted 2023-08-10; First posted 2023-08-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Acute Heart Failure
Keywords: Dapagliflozin; Acute heart failure; Decompensated heart failure; Hospitalization; Sodium-glucose cotransporter-2 inhibitors
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin group (Experimental): This group will receive oral Dapagliflozin 10 mg once daily within 24 hours from hospital admission, in addition to the standard treatment for acute heart failure.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Standard group (No Intervention): This group will only receive the standard treatment for acute heart failure.

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin is a drug that works through inhibition of sodium glucose transporter-2 resulting in glucosuria.
  Other Names: Sodium-glucose cotransporter-2 inhibitors
  Arms: Dapagliflozin group

SUMMARY:
The goal of this clinical trial is to evaluate the short-term clinical outcomes of starting Dapagliflozin on the same day of hospital admission in patients with acute decompensated heart failure (ADHF) with reduced ejection fraction.

The main questions it aims to answer are:

* Does early initiation of Dapagliflozin improve the length of hospital stay and in-hospital mortality in patients with ADHF?
* Does early initiation of Dapagliflozin enhance the diuretic response, weight reduction and pro-BNP reduction in the acute stage of HF?
* Does early initiation of Dapagliflozin adversely affect the hemodynamic stability and kidney functions in the acute stage of HF?

Participants will be randomized with the ratio of 1:1 within 24 hours of admission to receive Dapagliflozin 10 mg/day versus standard of care. Follow up will continue for 2 months after hospital discharge.

Researchers will compare the in-hospital and 60-day clinical outcomes in the Dapagliflozin group versus the standard treatment group.

DETAILED DESCRIPTION:
Background and Rationale:

With growing interest in studying the pharmacodynamics of SGLT-2 inhibitors, several cardio-protective mechanisms were defined beyond their diuretic effect. Those included anti-inflammatory effect and attenuation of oxidative stress in myocardial cells, renin-angiotensin aldosterone system blocking via activating AT-2 receptors, inhibition of Na+-H+ exchanger within myocardial cells , improving cardiac metabolomics via supplying more ketones , and weight reduction through lowering insulin secretion.

These findings invited more research to evaluate their benefit in patients having heart failure with reduced ejection fraction (HFrEF) regardless of diabetes mellitus (DM) status. Two large trials (DAPA-HF and EMPEROR-Reduced) have shown a consistent mortality benefit for SGLT-2 inhibitors in HFrEF patients in absence of DM.

Having a wide safety margin and low risk of complications, the use of SGLT-2 inhibitors was recently extended beyond the scope of cardiovascular disease to include patients with chronic kidney disease after their renal protective role was validated in CREDENCE and DAPA-CKD trials with significantly lower risk of albuminuria and disease progression.

Since most of the forementioned studies included patients with chronic HF who are stable on oral therapy, it has become urging to study the efficacy and safety of starting SGLT-2 inhibitors in patients with acute HF during the hospital phase. Ongoing trials have been investigating this issue recently, with pending outcomes. However, patients with de-novo AHF secondary to acute coronary syndrome have been excluded from these studies. Also, some of those studies started SGLT2 inhibitors only after stabilization of acute heart failure patients in-hospital.

Objectives:

The aim of this study is to evaluate the immediate and short-term clinical outcomes of starting Dapagliflozin in patients with acute decompensated heart failure with reduced ejection fraction during hospitalization.

Study Methods

* Population of study: Patients admitted to hospital with acute heart failure, either de-novo or acute decompensated on top of chronic.
* Study location: Kasr Al-Ainy Medical School, Cairo university.
* Recruitment location: Kasr Al-Ainy Medical School, Aswan Heart Centre.
* Methodology in details:

A-Full medical history including:

Age, gender, onset and duration of shortness of breath and NYHA functional class. Past history of DM, HTN, CAD, VHD, HF, stroke, other comorbidities, and smoking status will be obtained in all participants.

B-Full clinical examination including:

Assessment of body weight, height and calculation of BMI and BSA. Vital signs including blood pressure measurement using standard technique, assessment of the pulse, respiratory rate and temperature. Examination of all body systems.

C- Blood sample and chemistry:

Blood tests will be done to all participants. Lab workup will include CBC, liver and kidney function tests, electrolytes, HBA1C and lipid profile. Estimated GFR will be calculated using CKD-EPI equation.

D- Serum NT-proBNP:

On admission and on day 4 (or at discharge if earlier).

E- Electrocardiography (ECG):

12-lead ECG will be done for all participants. Data will be recorded including rhythm, ST-T changes, QRS width, and any form of conduction disturbance.

F- Conventional Transthoracic echocardiography (TTE):

TTE will be done for all patients on admission:

* Measure LV end-systolic and end-diastolic diameters.
* Measure LV systolic function by M-mode and Biplane Simpson's method.
* Measure LV diastolic function, E/A and E/e' ratio
* Calculate LA volume index.
* Calculate LV mass index.
* Assess cardiac valves (mitral, aortic and tricuspid valves).
* Estimate systolic pulmonary artery pressure.
* Measure RV dimensions and function.
* Measure RA area.

G. 2D-Speckle tracking echocardiography:

• Measure LV global longitudinal strain (GLS).

H. Randomization:

* Patients will be randomized with the ratio of 1:1 within 24 hours of admission to receive Dapagliflozin 10 mg/day versus standard of care (using online randomization https://en.calc-site.com/randoms/grouping). Treatment will continue for 2 months after discharge.
* Randomized treatment will be withheld in case of hypotension (SBP<90 mmHg), development of hypoglycemia < 80 mg/dl, metabolic acidosis, or >50% drop in eGFR for 2 consecutive measures.
* Randomized treatment will be resumed after resolution of the previously mentioned conditions.

I. Hospital course:

* Daily vital signs and assessment of fluid status.
* Daily fluid balance.
* Body weight change after 4 days of hospital admission or less if discharged earlier.
* Response to diuretics defined as adjusted urine output and adjusted weight change per 40 mg of IV furosemide or equivalent dose.
* Daily urea, creatinine and eGFR.
* Blood sugar monitoring.

J. Follow-up visits:

Patients will be followed in the outpatient clinic at 2 months after discharge, with the following data to be obtained:

1. NYHA class, and occurrence of any cardiac symptoms.
2. Need and reason for re-hospitalization.
3. History of dysuria, or genital discharge.
4. Medication intake and compliance.
5. Clinical examination including vital signs, body weight, and signs of left or right side HF.
6. Urea, creatinine and eGFR.
7. Electrolytes including Na and K.
8. HbA1C.

K. Follow-up serum NT-proBNP:

* At 2 months after discharge.
* Data will be compared to baseline values.

In case of mortality, data will be collected about the date and cause of mortality, and any reported clinical events before mortality.

* Potential risks:

  1. Mild pain during blood sample withdrawal.
  2. Low incidence of occurrence of side effects for Dapagliflozin including urinary tract infection, hypotension, and in rare cases hypoglycemia or metabolic acidosis.
* Confidentiality of data:

Data will be presented and used without inference to the name or personal data of the patients. All patient records will be handelled in accordance to hospital and national confidentiality protocols.

- Sample size :

Based on the results mentioned in a previously published similar study, where the frequency of composite endpoint of worsening HF, rehospitalization for HF or death at 60 days was 10% in the Empagliflozin group versus 33% in the placebo group, with a study power of 80% and a significance level of 5%, and by using an online sample size calculator (http://statulator.com/SampleSize/ss2P.html), the estimated sample size is 55 patients per group.

- Statistical analysis

Descriptive statistics will be summarized as mean ± SD for normally distributed continuous variables or otherwise as median and 25th to 75th percentile. Categorical variables will be described by frequencies and percentages. Differences in paired samples will be tested using the Wilcoxon signed-rank test or paired Student's t-test. Categorical variables will be compared using the chi-square or Fisher's exact test. Statistical significance is defined at a level of α ≤ 0.05.

Kaplan-Meier survival curves will be drawn to assess differences between groups for the time to an event. For the Cox model, univariate analysis of each of the possible predictors of the outcome will be tested, and only those variables that are significant at P<0.05 will be included in a multivariable model. A stepwise option will be used to determine independent predictors of the outcome variables.

Analysis will be performed with SPSS, Version 24 (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients above 18 years presenting with acute heart failure defined as rapid development of dyspnea NYHA class III-IV associated with clinical signs of HF (e.g. congested neck veins, pulmonary rales, lower limb swelling, radiological evidence of pulmonary congestion) with LVEF ≤ 40%.

Exclusion Criteria:

1. Cardiogenic shock on admission, defined as SBP < 90 mmHg plus signs of peripheral hypoperfusion or the need of vasopressor or inotropic support.
2. Estimated GFR < 30 mL/min/1.73 m2.
3. Pregnancy or lactation.
4. Type I DM or history of DKA.
5. Treatment with any SGLT2 inhibitor in the last month.
6. Known intolerance to any SGLT2 inhibitor.
7. Severe anemia (Hemoglobin < 7 g/dl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
All-cause mortality during hospitalization. | From the date of admission until the date of discharge, average of 7 days
  Death from any cause during the period of hospital stay.
Length of hospital stay | From the date of admission until the date of discharge, average of 7 days
  The number of days from hospital admission to discharge.
Diuretic response during the hospital phase. | First 4 days of hospital admission
  Defined as adjusted urine output and weight change per 40 mg of IV Furosemide or equivalent dose
Change in NT-proBNP at day 4 (or at discharge if earlier). | First 4 days of hospital admission
  The percentage change between baseline NT-proBNP on admission and NT-proBNP at day 4.

SECONDARY OUTCOMES:
Composite endpoint of cardiovascular death, re-admission for HF, or urgent clinic visit for decompensation at 2 months after hospital discharge. | 60 days after hospital discharge
  Decompensation is defined as worsening symptoms +/- signs of HF requiring intensification of diuretic dose.
Change in serum NT-proBNP after 2 months. | 60 days after hospital discharge
  The percentage change between baseline NT-proBNP and 2 months after discharge.
Worsening renal functions | During hospital stay and up to 60 days after hospital discharge
  Defined as > 50% worsening of baseline eGFR, or absolute drop below 30 ml/min/1.73 m2.
Composite endpoint of urogenital infections, hypoglycemic events, hypotension events or diabetic ketoacidosis. | During hospital stay and up to 60 days after hospital discharge
  Reporting any side effects that could be due to Dapagliflozin after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Abdelhamid, Professor, Principal Investigator — Chairman of Cardiology Department, Cairo University
Locations (2):
- Egypt (2):
  - Aswan Heart Centre, Aswān
  - Kasr Al-Ainy Medical School, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest. Data or samples shared will be coded, with no reference to participants' identity.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan.

REFERENCES:
- [Background] Damman K, Beusekamp JC, Boorsma EM, Swart HP, Smilde TDJ, Elvan A, van Eck JWM, Heerspink HJL, Voors AA. Randomized, double-blind, placebo-controlled, multicentre pilot study on the effects of empagliflozin on clinical outcomes in patients with acute decompensated heart failure (EMPA-RESPONSE-AHF). Eur J Heart Fail. 2020 Apr;22(4):713-722. doi: 10.1002/ejhf.1713. Epub 2020 Jan 7. PMID 31912605
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Ul Amin N, Sabir F, Amin T, Sarfraz Z, Sarfraz A, Robles-Velasco K, Cherrez-Ojeda I. SGLT2 Inhibitors in Acute Heart Failure: A Meta-Analysis of Randomized Controlled Trials. Healthcare (Basel). 2022 Nov 23;10(12):2356. doi: 10.3390/healthcare10122356. PMID 36553880